CLINICAL TRIAL: NCT04759014
Title: The Effect of Using Two Different Prosthetic Feet on Functional Capacity, Pain Severity, Satisfaction Level and Quality of Life in High Activity Patients With Unilateral Transtibial Amputation
Brief Title: The Effect of Using Two Different Prosthetic Feet in Patients With Unilateral Transtibial Amputation
Status: Completed | Type: Observational
Sponsor: Gaziler Physical Medicine and Rehabilitation Education and Research Hospital (Other)
Responsible Party: Principal Investigator, Yasin Demir, Physical Medicine and Rehabilitation Associate Professor, Gaziler Physical Medicine and Rehabilitation Education and Research Hospital
Other Study IDs: 11
Record Dates: First submitted 2021-02-13; First posted 2021-02-17 (Actual); Last update posted 2021-11-23 (Actual); Status verified 2021-11

CONDITIONS: Amputation
Keywords: Transtibial amputation; Prosthetic foot; Functional capacity; Satisfaction; Quality of life
MeSH Terms: conditions — Personal Satisfaction | interventions — Quality of Life

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group 1: 21 patients using non-articulated dynamic foot (non-articulating ankle, NAA)
  Interventions: Other: The effect of using two different prosthetic feet on functional capacity, pain severity, satisfaction level and quality of life
- Group 2: 21 patients using dynamic foot with hydraulic ankle (articulating hydraulic ankle, AHA)
  Interventions: Other: The effect of using two different prosthetic feet on functional capacity, pain severity, satisfaction level and quality of life

INTERVENTIONS:
Other: The effect of using two different prosthetic feet on functional capacity, pain severity, satisfaction level and quality of life — The effect of using two different prosthetic feet on functional capacity, pain severity, satisfaction level and quality of life

SUMMARY:
Background: Prescribing optimal prosthetic feet to ensure successful rehabilitation is difficult since there are no generally established clinical guidelines based on objective data.

Aim: To investigate the effect of using non-articulated dynamic foot (non-articulating ankle, NAA) and dynamic foot with hydraulic ankle (articulating hydraulic ankle, AHA) on functional capacity, pain severity, satisfaction level and quality of life (QoL) in high activity patients with unilateral transtibial amputation.

DETAILED DESCRIPTION:
Background: Prescribing optimal prosthetic feet to ensure successful rehabilitation is difficult since there are no generally established clinical guidelines based on objective data.

Aim: To investigate the effect of using non-articulated dynamic foot (non-articulating ankle, NAA) and dynamic foot with hydraulic ankle (articulating hydraulic ankle, AHA) on functional capacity, pain severity, satisfaction level and quality of life (QoL) in high activity patients with unilateral transtibial amputation.

Methods: Forty-two patients with unilateral transtibial traumatic amputation will be participated in this cross-sectional study. Functional capacity will be evaluated using the six-minute walking test (6MWT). The severity of residual limb pain, sound limb pain and low back pain will be evaluated with a 10-point Visual Analogue Scale (VAS). The socket system, prosthetic foot and overall prosthesis satisfaction will be evaluated with a 10-point VAS. The QoL of each patient will be assessed using the Short Form 36 (SF-36).

ELIGIBILITY:
Inclusion Criteria:

* aged 18-65 years
* Medicare functional classification level K4 (very active)
* using the prosthesis for at least 6 months and at least 6 hrs a day
* using active vacuum-assisted suspension system

Exclusion Criteria:

* bilateral amputation,
* the presence of neurological, cardiovascular and pulmonary disease that could affect walking performance.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Fourty-two patients with unilateral transtibial traumatic amputation will be participated in this cross-sectional study. Only participants using active vacuum-assisted suspension system will be included in the study in order to prevent any bias from suspansion system on the results.
Sampling Method: Non-Probability Sample
Enrollment: 42 (Actual)
Dates: Start 2021-02-18 (Actual); Primary Completion 2021-07-01 (Actual); Study Completion 2021-07-01 (Actual)

PRIMARY OUTCOMES:
Visual Analogue Scale | through study completion, an average of one and a half months
  All patients will mark the severity of residual limb pain, sound limb pain and low back pain on a Visual Analogue Scale (VAS; from 0 (no pain) to 10 (worst pain)). The socket system, prosthetic foot and overall prosthesis satisfaction will be evaluated with a 10-point VAS (from 0 (absolutely dissatisfied) to 10 (absolutely satisfied)).
Short Form 36 (SF-36) | through study completion, an average of one and a half months
  The QoL of each patient will be assessed using the Short Form 36 (SF-36). The validity and reliability of the Turkish version of SF-36 has been demonstrated. SF-36 consists of 36 questions on eight different subscales that include physical functioning, role limitations due to physical health problems, bodily pain, general health perceptions, energy and fatigue, vitality, social functioning, role limitations due to emotional problems and general mental health. Each subscale of SF-36 is scored between 0 and 100, and higher scores illustrate better QoL.
The six-minute walking test (6MWT) | through study completion, an average of one and a half months
  Functional capacity will be evaluated using the six-minute walking test (6MWT). The 6MWT evaluates walking function and endurance. Patients will be instructed to walk quickly, safely, and as much distance as possible along a rectangular path. The 6MWT is both valid and reliable among individuals with lower-limb loss.

SECONDARY OUTCOMES:
Likert scale | through study completion, an average of one and a half months
  Level of difficulty experienced during walking on straight road, walking uneven road, ascending stairs, descending stairs, ascending ramps and descending ramps will be recorded on a 5-point Likert scale ((1) very easy, (2) easy , (3) neutral, (4) difficult, (5) very difficult).

CONTACTS AND LOCATIONS:
Overall Officials: Merve Orucu Atar, MD, Principal Investigator — Gaziler Physical Medicine and Rehabilitation, Training and Research Hospital, Department of PMR
Locations (1):
- Gaziler Physical Medicine and Rehabilitation, Education and Research Hospital, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No